CLINICAL TRIAL: NCT01579838
Title: An Open Label Study of the Effects of Eculizumab in CD59 Deficiency
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hadassah Medical Organization (Other)
Responsible Party: Principal Investigator, Mevorach Dror, Head of Medicine and head of Rheumatology Research Center, Hadassah Medical Organization
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CD59-Mevorach-1
Record Dates: First submitted 2012-02-23; First posted 2012-04-18 (Estimated); Last update posted 2012-04-18 (Estimated); Status verified 2012-04

CONDITIONS: Chronic Hemolysis
MeSH Terms: interventions — eculizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Eculizumab (Experimental): Eculizumab will be administrated according to known protocols.
  Interventions: Drug: Eculizumab

INTERVENTIONS:
Drug: Eculizumab — PNH and or atypical TTP classical protocols
  Other Names: Soliris

SUMMARY:
The investigators have identified patients with CD59 deficiency that suffers from chronic hemolysis and peripheral demyelinating disease. It was shown that complement terminal pathway can cause inflammation in the peripheral nervous system. Complement can greatly increase the immune attack in the nerves. Eculizumab has already been shown to be effective in a rare blood disorder known as paroxysmal nocturnal hemoglobinuria (PNH). Attacks of PNH are also mediated through complement. Therefore, the investigators of this study are investigating whether by 'turning off' complement in CD59 deficiency, further attacks of hemolysis and nerve injury can be avoided and whether the neurological status will ameliorate.

DETAILED DESCRIPTION:
It has been shown in some scientific studies that lack of CD59 in the context of the disease paroxysmal nocturnal hemoglobinuria (PNH)leads to chronic hemolysis. The investigators have identified patients wirh CD59 deficiency that suffers from chronic hemolysis and demyelinating disease. It was shown that complement terminal pathway can cause cause inflammation in nervous system. Complement can greatly increase the immune attack in the nerves. Eculizumab has already been shown to be effective in a rare blood disorder known as PNH. Attacks of PNH are also mediated through complement. Therefore, the investigators of this study are investigating whether by 'turning off' complement in CD59 deficiency, further attacks of hemolysis and nerve injury can be avoided.

The primary (most important) objectives of this study are to determine:

Whether Eculizumab ameliorate the neurological condition documented in the last month before treatment and whether it reduces the relapse frequency in patients with relapsing chronic inflammatory demyilinating polyneuropathy. The number of attacks during the one year treatment period will be compared to the number of attacks that occurred prior to initiation of eculizumab treatment. For patients with more than 2 year disease duration, the average number of attacks in the preceding 2 years will be calculated. For patients with less than 2 years disease duration the number of attacks in the preceding year will be used.

Whether Eculizumab reduces chronic hemolysis as judged by LDH levels, and haptoglobin, and level of hemoglobin. the same for corticosteroids and or I.V. IgG consumption before and after treatment with eculizumab.

The safety profile of eculizumab in patients with CD59 deficiency will be determined by parents report evry other week, documentation of clinic referral and hospitalizations. The number of participants with advers events will be determined.

The secondary objectives are to determine:

Whether eculizumab maintains or improves limbs motion, function and quality of life as measured by a variety of established disability scales like the modified SF36 and like a questionaire developed for this age group. The investigators will also assess the severity of an individual attack and the degree of recovery.

How the drug behaves in the patient's blood by measuring the presence of membrane attack complex on neutrophils and red blood cells.

ELIGIBILITY:
Inclusion Criteria:

* CD59 deficiency

Exclusion Criteria:

* recent exposure to meningococcal infections

Ages: 2 Months to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 5 (Estimated)
Dates: Start 2012-02; Primary Completion 2013-03 (Estimated); Study Completion 2013-03 (Estimated)

PRIMARY OUTCOMES:
Whether Eculizumab reduces chronic hemolysis | 8 months
  The primary objectives of this study are to determine:
  Whether Eculizumab reduces chronic hemolysis as judged by LDH levels, and haptoglobin, and level of hemoglobin.
Steroid and iv IgG cumulative dosage | 8 months
  Cumulative steroid and IgG dosage before and after treatment
Safety. | 8 months
  Whether the subjects develop known or possible related side effect to the treatment. The number of participants that develop adverse effects will be determined. reports from parents will be taken avery other week and documented clini or hospital visits will be included.
Whether Eculizumab ameliorates the neurological status compared to one month before treatment | 8 months
  The neurological status in the last month prior to treatment will be determined followed by neurological staus examination every two weeks.

SECONDARY OUTCOMES:
Whether eculizumab maintains or improves limbs motion | 8 months
  Whether there is a neurological amelioration
function and quality of life as measured by a variety of established disability scales. | 8 months
  we will be using evry other week parents report of his clinical condition. We will use modified SF36 and local questionairre.
The severity of an individual attack and the degree of recovery. | 8 months
Levels of membrane attack complex | 8 months
  This will be measured using flow cytometry for the presence of membrane attack complex on neutrophild and res blood cells.

CONTACTS AND LOCATIONS:
Overall Officials: Dror Mevorach, MD, Principal Investigator — hmo
Locations (1):
- Hadassah Medical Center, Jerusalem, Israel

REFERENCES:
- [Derived] Mevorach D, Reiner I, Grau A, Ilan U, Berkun Y, Ta-Shma A, Elpeleg O, Shorer Z, Edvardson S, Tabib A. Therapy with eculizumab for patients with CD59 p.Cys89Tyr mutation. Ann Neurol. 2016 Nov;80(5):708-717. doi: 10.1002/ana.24770. Epub 2016 Sep 19. PMID 27568864